CLINICAL TRIAL: NCT06276998
Title: A Randomized Double-Blind Placebo-controlled Phase Ⅲ Clinical Trial Evaluating the Efficacy and Safety of LNK01001 (Zemprocitinib) in Patient With Moderate-to-Severe Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Biologic Disease-Modifying Antirheumatic Drugs (COURAGE-RA)
Brief Title: A Study of LNK01001 Capsule in Subjects With Active Rheumatoid Arthritis (COURAGE-RA)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lynk Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LK001304
Record Dates: First submitted 2024-02-02; First posted 2024-02-26 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LNK01001 12 mg (Experimental): Period 1: Participants receive LNK01001 12 mg twice daily for 24 weeks. Period 2: Participants will continue on LNK01001 12 mg twice daily from Week 24 to Week 76.
  Interventions: Drug: LNK01001
- Placebo / LNK01001 12 mg (Placebo Comparator): Period 1: Participants receive a placebo twice daily for 24 weeks. Period 2: Participants will switch to receive LNK01001 12 mg twice daily from Week 24 to Week 76.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LNK01001 — Capsule; Oral
  Arms: LNK01001 12 mg
Drug: Placebo — Capsule; Oral
  Arms: Placebo / LNK01001 12 mg

SUMMARY:
Brief Summary: This is a randomized, double-blind study comparing LNK01001 to placebo in Chinese participants with moderately to severely active rheumatoid arthritis who are on a stable dose of conventional synthetic disease-modifying anti-rheumatic drugs (csDMARDs) and have an inadequate response or Intolerance to biologic DMARDs(bDMARDs).

The study objective of Period 1 (Day 1 to Week 24) is to compare the safety and efficacy of LNK01001 12 mg twice daily (BID) versus placebo for the treatment of signs and symptoms of participants with moderately to severely active rheumatoid arthritis (RA) who are on a stable dose of csDMARDs and had an inadequate response to or intolerance to at least 1 bDMARD.

The study objective of Period 2 (Week 24 to Week 76) is to evaluate the long-term safety, tolerability, and efficacy of LNK01001 12 mg BID in participants with RA who completed Period 1.

DETAILED DESCRIPTION:
This study includes a 35-day screening period; a 24-week randomized, double-blind, parallel-group, placebo-controlled treatment period (Period 1); a 52-week open label long-term extension period (Period 2); and a 28 to 35-day follow-up period (FU).

Participants who meet eligibility criteria will be randomized in a 1:1 ratio to two treatment groups:

Group 1: LNK01001 12 mg BID (Day 1 to Week 24)， LNK01001 12 mg BID (Week 24 and thereafter)

Group 2: Placebo (Day 1 to Week 24)， LNK01001 12 mg BID (Week 24 and thereafter)

Participants who complete the Week 24 visit (end of Period 1) will enter the extension portion of the study, Period 2, and continue to receive LNK01001 12 mg BID treatment. Starting at Week 12, rescue therapy is allowed if there's less than 20% improvement in both swollen joint count (SJC) and tender joint count (TJC) compared to Baseline. Starting at Week 24, initiation of or change in corticosteroids, non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen, or adding or increasing doses in up to 2 csDMARDs (concomitant use of up to 2 csDMARDs except the combination of methotrexate and leflunomide) is allowed.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 and above.
* Diagnosis of rheumatoid arthritis (RA) for ≥ 3 months.
* ≥ 6 swollen joints (based on 66 joint counts) and ≥ 6 tender joints (based on 68 joint counts) at Screening and baseline visit.
* Erythrocyte sedimentation rate (ESR) ≥ 28mm/h or high-sensitivity C-Reactive Protein (hsCRP) ≥ ULN at Screening.
* Participants have been receiving csDMARD therapy ≥ 3 months and on a stable dose for ≥ 4 weeks prior to the first dose of study drug.
* Have an inadequate response to ≥ 1 bDMARD.

Exclusion Criteria:

* Subjects who were prior exposure to Janus Kinase (JAK) inhibitor (including but not limited to tofacitinib, baricitinib, and filgotinib) and have evidence showing an inadequate response or intolerance.
* Subjects who received intra-articular, intramuscular, intravenous, trigger point or tender point, intracapsular, or intra-tendon injections of glucocorticoids within 4 weeks before randomization.
* Current diagnosis of systemic inflammatory disease other than RA.
* History of malignancy or current diagnosis of malignancy within 5 years before screening visit.
* Uncontrolled diabetes, hypertension, kidney disease, liver disease, severe heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 24 | Baseline and Week 24
  Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR20 response criteria:
  1. 20% improvement in 68-tender joint count;
  2. 20% improvement in 66-swollen joint count; and
  3. 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).

SECONDARY OUTCOMES:
Change from Baseline in Disease Activity Score 28 (DAS28) (CRP) at week 24 | Baseline and Week 24
  The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
Percentage of Participants with an American College of Rheumatology 50% (ACR50) Response at week 24 | Baseline and Week 24
  Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR50 response criteria:
  1.50% improvement in 68-tender joint count; 2.50% improvement in 66-swollen joint count; and 3.50% improvement in at least 3 of the 5 following parameters:
  * Physician global assessment of disease activity
  * Patient global assessment of disease activity
  * Patient assessment of pain
  * Health Assessment Questionnaire - Disability Index (HAQ-DI)
  * High-sensitivity C-reactive protein (hsCRP).
Change from Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) at all visits. | Baseline to Week 76.
  The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. A negative change from Baseline in the overall score indicates improvement.
Percentage of Participants with an American College of Rheumatology 70% (ACR70) Response at all visits. | Baseline to Week 76.
  Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR70 response criteria:
  1. 70% improvement in 68-tender joint count;
  2. 70% improvement in 66-swollen joint count; and 3.70% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Percentage of Participants Achieving Low Disease Activity (LDA) Based on DAS28(CRP) at all visits. | Baseline to Week 76.
  Low disease activity. was defined as a DAS28 score less than or equal to 3.2.The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
Percentage of Participants Achieving Clinical Remission (CR) Based on DAS28(CRP) at all visits | Baseline to Week 76.
  Clinical remission was defined as a DAS28 (CRP) score less than 2.6.The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
Percentage of Participants with an American College of Rheumatology 20% (ACR20) Response at all visits (except week 24). | Baseline to Week 76 (except week 24).
  Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR20 response criteria:
  1.20% improvement in 68-tender joint count; 2. 20% improvement in 66-swollen joint count; and 3. 20% improvement in at least 3 of the 5 following parameters:
  * Physician global assessment of disease activity
  * Patient global assessment of disease activity
  * Patient assessment of pain
  * Health Assessment Questionnaire - Disability Index (HAQ-DI)
  * High-sensitivity C-reactive protein (hsCRP).
Change from Baseline in the Severity of Morning Stiffness at all visits. | Baseline to Week 76.
  Morning stiffness severity was determined by the Patient's Assessment of Severity and Duration of Morning Stiffness questionnaire. Participants rated the severity of morning stiffness on awakening over the past 7 days on a scale from 0 (No morning stiffness) to 10 (Worst possible morning stiffness).

CONTACTS AND LOCATIONS:
Overall Officials: Linda Wei, Study Director — Lynk Pharmaceuticals
Locations (1):
- Peking Union Medical College Hospital, Beijing, China